CLINICAL TRIAL: NCT01369485
Title: Multi-center, Prospective, Randomized, Double-blind, Sham-controlled Clinical Study to Evaluate Safety and Effectiveness of a Transcutaneous, High-frequency, Amplitude-modulated, Non-invasive Neuromodulation Device on Urgency Urinary Incontinence in Subjects With Overactive Bladder (OAB)
Brief Title: Safety and Effectiveness of a Non-invasive Neuromodulation Device on Urgency Urinary Incontinence in Overactive Bladder
Acronym: Beacon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ethicon Endo-Surgery (Industry)
Collaborators: Novella Clinical (Other); Data & Inference, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CI-10-0009
Record Dates: First submitted 2011-05-24; First posted 2011-06-09 (Estimated); Results first posted 2014-09-11 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Overactive Bladder
Keywords: Urinary Incontinence; Overactive Bladder; Frequency; Urgency
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Treatment group (Active Comparator): VERV™ System
  Interventions: Device: (VERV™ System)
- Sham Treatment Group (Sham Comparator): Sham version of (VERV™ System)
  Interventions: Device: Sham version of (VERV™ System)

INTERVENTIONS:
Device: (VERV™ System) — Active electrode patches are worn for 12 weeks, one per week. The patch is placed by the subject. All subjects will have access to active patches for 9 months after the sham-controlled 12-week portion of the study is complete.
  Other Names: Non-invasive neurostimulation device
  Arms: Active Treatment group
Device: Sham version of (VERV™ System) — Inactive (sham) electrode patches are worn for 12 weeks, one per week. The patch is placed by the subject. All subjects will have access to active patches for 9 months after the sham-controlled 12-week portion of the study is complete.
  Other Names: Inactive Non-invasive neurostimulation device
  Arms: Sham Treatment Group

SUMMARY:
The purpose of this study is to evaluate the change from baseline between the active and sham treatment groups in the treatment of urgency (urinary) incontinence episodes (leaks).

ELIGIBILITY:
Inclusion Criteria:

* Males and Females, at least 18 years of age
* Failure on primary OAB treatment, such as behavior modification or fluid/diet management, AND at least one (1) anti-cholinergic drug (unless patient was contra-indicated for anti-cholinergic use)
* Symptoms of overactive bladder for at least 6 months
* An average of one (1) or more urgency (urinary) incontinence episodes per 24-hours, over a 3-day period, confirmed by the 3-day baseline voiding diary, with a maximum of 12 urgency (urinary) incontinence episodes per 24-hours
* Dexterity and ability to place and operate the device
* Females of child-bearing capability agrees to use a reliable form of birth control for the duration of the trial
* An average of eight (8) or more voids per 24-hours, over a 3-day period, confirmed by the 3-day baseline voiding diary
* Willing and capable of understanding and complying with all requirements of the protocol, including proper completion of the baseline voiding diary
* Signed and dated the IRB-approved Informed Consent document.

Exclusion Criteria:

* Dysfunctional voiding symptoms unrelated to OAB, such as clinically significant bladder outlet obstruction, and urinary retention (pvr > 100 cc)
* Morbidly obese, defined as having Body Mass Index (BMI) > 40 kg/m2
* Stress predominant mixed urinary incontinence
* Neurological disease affecting urinary bladder function, including but not limited to Parkinson's disease, multiple sclerosis, stroke, spinal cord injury and uncontrolled epilepsy.
* Pelvic surgery (such as sub-urethral sling, pelvic floor repair) within the past 6 months
* Intravesical or urethral sphincter Botulinum Toxin Type A injections within the past 12 months
* Any neuromodulation therapy for overactive bladder within the past 3 months
* Failure to respond to previous neuromodulation therapy for overactive bladder
* Leading edge of any vaginal prolapse is beyond hymenel ring.
* Prior peri-urethral or transurethral bulking agent injections for bladder problems within the past 12 months.
* Any skin conditions affecting treatment or assessment of the treatment sites
* History of lower back surgery or injury that could impact placement of the patch, or where underlying scar tissue or nerve damage may impact treatment.
* Presence of an implanted electro-medical device (e.g. pacemaker, defibrillator, InterStim®, etc.), or any metallic implant in the lower back.
* Pregnant, nursing, suspected to be pregnant (by urine pregnancy method), or plans to become pregnant during the course of the study.
* Known latex allergies, or allergies or hypersensitivity to patch materials that will be in contact with the body (e.g., hydrogel, acrylic-based adhesive, polyurethane).
* Uncontrolled diabetes and/or diabetes with peripheral neuropathy.
* Current Urinary Tract Infection (UTI) or history of recurrent UTIs (>3 UTIs in the past year).
* History of lower tract genitourinary malignancies within the last 6 months or any previous pelvic radiation.
* Any clinically significant systemic disease or condition that in the opinion of the Investigator would make the patient unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2011-06; Primary Completion 2013-01 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kennelly, MD, Principal Investigator — McKay Urology
Locations (14):
- United States (14):
  - Arizona Urologic Specialists, Tucson, Arizona
  - Tri Valley Urology Medical Group, Murrieta, California
  - GW Medical Faculty Associates, Washington D.C., District of Columbia
  - Specialists in Urology, Naples, Florida
  - Urology Center of Florida, Pompano Beach, Florida
  - Women's Health Institute of Illlinois, Ltd, Oak Lawn, Illinois
  - 1st Urology, PSC dba Metropolitan Urology, Jeffersonville, Indiana
  - William Beaumont Hospital, Royal Oak, Michigan
  - University Urology Associates, New York, New York
  - McKay Urology, Charlotte, North Carolina
  - Alliance Urology Specialists, P.A., Greensboro, North Carolina
  - Carolina Urologic Research, Myrtle Beach, South Carolina
  - Integrity Medical Research, Mountlake Terrace, Washington
  - Wheaton Franciscan Medical Group - Milwaukee Urogynecology, Wauwatosa, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After informed consent was obtained, subjects had a 10-day washout period from any anti-cholinergic medications prescribed for treatment of overactive bladder prior to initiating study treatment.
Groups:
- Randomized Active Treatment Group: VERV™ System
  (VERV™ System): Active electrode patches are worn for 12 weeks, one per week. The patch is placed by the subject. All subjects will have access to active patches for 9 months after the sham-controlled 12-week portion of the study is complete.
  Patients completing ther randomized phase of the study were rolled over to receive active treatment with VERV™ System for up to 9 additional months.
- Randomized Sham Treatment Group: Sham version of (VERV™ System)
  Sham version of (VERV™ System): Inactive (sham) electrode patches are worn for 12 weeks, one per week. The patch is placed by the subject. All subjects will have access to active patches for 9 months after the sham-controlled 12-week portion of the study is complete.
  Patients completing ther randomized phase of the study were rolled over to receive active treatment with VERV™ System for up to 9 additional months.
Period: Randomized Phase (Day 0 to Week 12)
Arm/Group | Randomized Active Treatment Group | Randomized Sham Treatment Group
Started | 80 | 83
Completed | 57 | 66
Not Completed | 23 | 17
Not completed — Adverse Event | 7 | 5
Not completed — Withdrawal by Subject | 12 | 8
Not completed — Lost to Follow-up | 2 | 4
Not completed — expired patches | 2 | 0
Period: Open Label Phase (Week 12 to Month 12)
Arm/Group | Randomized Active Treatment Group | Randomized Sham Treatment Group
Started | 57 | 66
Completed | 24 | 26
Not Completed | 33 | 40
Not completed — Adverse Event | 11 | 9
Not completed — Lost to Follow-up | 2 | 3
Not completed — Physician Decision | 3 | 4
Not completed — Withdrawal by Subject | 17 | 20
Not completed — Death | 0 | 1
Not completed — 1 pacemaker, 1 noncompliance, 1 hospice | 0 | 3

BASELINE CHARACTERISTICS:
Population: Intent to treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Treatment Group | Sham Treatment Group | Total
Number analyzed (Participants) | 80 | 83 | 163
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (14.3) | 62.4 (13.8) | 61.6 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 68 | 138
  Male | 10 | 15 | 25
Race/Ethnicity, Customized [Number; unit: participants]
  Native American | 1 | 1 | 2
  Asian | 1 | 2 | 3
  African American | 11 | 12 | 23
  Caucasian | 65 | 66 | 131
  Other | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 80 | 83 | 163

OUTCOME MEASURES:

1. Primary Outcome: Evaluate Proportion of Responders Based on the Change From Baseline in Mean Urgency (Urinary) Incontinence Episodes (Leaks) Between the Active and Sham Treatment Groups
Description: The primary objective of the randomized phase of the study is to evaluate the 12 week change from baseline in mean urgency (urinary) incontinence episodes (leaks) between the active and sham treatment groups. The mean of the number of urinary incontinence episodes over 24 hours" is defined as the mean of the number of UIEs recorded per 24 hour period for three consecutive days (via a 3-day diary).
  The primary objective of the open label phase of the study is to evaluate and confirm the continued efficacy of the VERV™ System for long-term use. The primary objective was assessed with rate of responders, where responder was defined as a subject who achieved a decrease of ≥50% in mean urgency urinary incontinence episodes at 12 weeks compared to baseline.
Time Frame: 12 weeks (Randomized Phase) and 12 Months (Open Label)
Population: Intent to treat population. Responders are defined as patients who had a greater than or equal to 50% decrease in mean number urgency incontinence episodes over 24 hours.
Measure: Number; unit: Number of responders
Groups:
- Open Label Active Treatment Group; Open Label Sham Treatment Group: Patients received active treatment with the VERV™ System for up to 9 additional months as part of the open label phase of the study.
Arm/Group | Active Treatment Group | Sham Treatment Group | Open Label Active Treatment Group | Open Label Sham Treatment Group
Number analyzed (Participants) | 80 | 83 | 25 | 26
Number of responders | 31 (3.03) | 38 (2.79) | 16 | 19
Statistical Analysis 1: Comparison: Active Treatment Group vs Sham Treatment Group; The sample size calculation was determined using the 2-sided Chi-square test with a significance level of 5% and 80% power based upon the following assumptions: (1) proportion of responders at end of 12 weeks of treatment would be 50% in the active (test) group and 25% in the inactive (control) group; (2) a responder was defined as a subject who experienced decrease of ≥50% in mean urgency urinary incontinence episodes (leaks) between baseline and Week 12 of the study; (3) 20 % dropout rate; Test type: Superiority or Other; p = 0.3636, Chi-squared
Statistical Analysis 2: Comparison: Open Label Active Treatment Group vs Open Label Sham Treatment Group; Test type: Superiority or Other; p = 0.4849, Chi-squared

2. Secondary Outcome: Measure Change in the Median of the Mean Urinary Frequency
Description: Evaluate the 12 week change from baseline in median urinary frequency between the active and sham treatment groups.
  Mean urinary frequency episodes calculated for each patient during time period. The median change in frequency was then calculated for each treatment group. Distribution of changes from baseline were then assessed prospectively for normality using the Kolmogorov - Smirnoff test. Since departure from normality was actually observed in the distribution, the Wilcoxon Rank-Sum test was performed to compare the median change between treatment groups and the p-values for the test of equality of medians were reported along with the medians.
Time Frame: 12 weeks and 12 Months
Measure: Median (Inter-Quartile Range); unit: Episodes/24 hours
Groups:
- Open Label Treatment Group; Open Label Sham Treatment Group: VERV™ System
  (VERV™ System): Active electrode patches are worn for 12 weeks, one per week. The patch is placed by the subject. All subjects will have access to active patches for 9 months after the sham-controlled 12-week portion of the study is complete.
Arm/Group | Active Treatment Group | Sham Treatment Group | Open Label Treatment Group | Open Label Sham Treatment Group
Number analyzed (Participants) | 80 | 83 | 25 | 26
Episodes/24 hours | -1.0 (3.07) [-2.7 to 0.3] | -1.3 (2.91) [-3.0 to -0.3] | -1.0 [-3.3 to 0.3] | -2.8 [-4.3 to 0.0]
Statistical Analysis 1: Comparison: Active Treatment Group vs Sham Treatment Group; Test type: Superiority or Other; p = 0.2893, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Open Label Treatment Group vs Open Label Sham Treatment Group; Test type: Superiority or Other; p = 0.3223, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Measure Median Change in Mean Volume Per Void
Description: Evaluate the 12 week median change from baseline in mean volume (ml) per void between the active and sham treatment groups
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: ml
Arm/Group | Active Treatment Group | Sham Treatment Group
Number analyzed (Participants) | 80 | 83
ml | 1.0 (50.20) [-26.6 to 23.5] | 8.8 (51.43) [-24.3 to 33.3]
Statistical Analysis 1: Comparison: Active Treatment Group vs Sham Treatment Group; Test type: Superiority or Other; p = 0.3387, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Measure Decrease in the Median Change From Baseline in Mean Urgency Episodes
Description: Evaluate the 12 week change from baseline in median for mean number of urgency episodes between the active and sham treatment groups.
  Patients were required to complete seven 3-day voiding diaries throughout the course of the study. The voiding diary collected the following information: amount voided (in ml); urgency associated with each toileted void , approximate time of leak, and presence of urge preceding leak.The mean number of urgency episodes over 24 hours was then calculated for each patient during the observation period. The change in median for the mean of the number of urgency episodes over 24 hours) for each treatment group was then calculated.
  Distribution of changes from baseline were assessed prospectively using the Kolmogorov - Smirnoff test. The Wilcoxon Rank-Sum test was performed to compare the median change between treatment groups and the p-values for the test of equality of medians were reported along with the medians.
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: Difference in episodes/24 Hours
Arm/Group | Active Treatment Group | Sham Treatment Group
Number analyzed (Participants) | 80 | 83
Difference in episodes/24 Hours | -1.7 (3.08) [-3.3 to 0.3] | -1.7 (3.32) [-3.3 to -0.3]
Statistical Analysis 1: Comparison: Active Treatment Group vs Sham Treatment Group; Test type: Superiority or Other; p = 0.6557, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Measure Improvement in the Median of the Mean OAB-Symptom Composite Score
Description: OAB Symptom Composite Score (OAB-SCS) is a composite symptom score of toilet voids, urgency severity and urge urinary incontinence combining the Indevus Urgency Severity Scale (IUSS) for capture of urgency severity per toilet void with 24-hour frequency and UUI episodes.
  IUSS Score/void and/or UUI is assigned an OAB-SCS Point/Void: 0(none)=1, 1(mild/easily tolerated)=2, 2(moderate discomfort interfering with activities)=3, 3(severe/extreme urgency discomfort that abruptly stopped all activity or tasks)=4, UUI without void=5.
  Overall OAB-SCS Score is calculated for each day by multiplying the OAB-SCS Points/Void and/or UUIs by the number of events meeting criteria and adding the individual scores together. The minimum overall OAB-SCS score in a 24 hour period would be a 1 (representing a single mild void with a OAB -SCS Point/Void score of 0). The score would increase based upon the number voids/events and overall severity each event. Medians calculated for each treatment group.
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Active Treatment Group | Sham Treatment Group
Number analyzed (Participants) | 80 | 83
units on a scale | -5.8 (16.46) [-14.7 to 1.3] | -8.0 (15.67) [-15.3 to 0.3]
Statistical Analysis 1: Comparison: Active Treatment Group vs Sham Treatment Group; Test type: Superiority or Other; p = 0.4354, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change in Median Total Health Related Quality of Life (HRQL) of OAB-q From Baseline (Screening) to Week 12
Description: The OAB-q is validated to measure symptom bother and life impact due to OAB. It consists of an 8-item Bother Scale to assess individual symptoms and a 25-item HRQL scale that in turn consists of 4 subscales (coping-8 items, concern-7 items, sleep-5 items and social-5 items) to assess impact on life. Responses for each item in the Bother Scale range from 1 (bothered not at all by the symptom) to 6 (Bothered A Very Great Deal). Scores are then added generating an overall Bother Score (severity) ranging from 8 to 48. For HRQL, individual responses range between 1-None of the Time to a 6-All of the Time. Subscale scores range from 8-48 (coping) 7-42 (concern), 5-30 (sleep) and 5-30 (social). Subscale scores are then added to generate the HRQL ranging between 25-150. Raw HRQL scores are transformed for standardization purposes as follows: ((Highest Possible Score-Actual Raw Score)/Range of Scores)*1 00 so that scores could range from 0 (All of the Time) to 100 (None of the Time).
Time Frame: 12 Weeks (Randomized Phase) and 12 Months (Open Label).
Population: Intent to Treat
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Active Treatment Group | Sham Treatment Group | Open Label Active Treatment Group. | Open Label Sham Treatment Group
Number analyzed (Participants) | 56 | 66 | 25 | 28
units on a scale | 8.8 (20.28) [1.6 to 20.0] | 9.2 (22.05) [-0.8 to 27.2] | 19.2 (23.88) [2.4 to 28.8] | 24.0 (20.30) [9.2 to 32.4]
Statistical Analysis 1: Comparison: Active Treatment Group vs Sham Treatment Group; Test type: Superiority or Other; p = 0.9918, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Open Label Active Treatment Group. vs Open Label Sham Treatment Group; Test type: Superiority or Other; p = 0.3770, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Change in Patient Perception of Bladder Condition (PPBC) From Baseline (Screening Period) to Week 12 as Defined as an Improvement in Severity.
Description: PPBC is a 6-point scale (from 'no problems at all' to 'many severe problems') describing the problem level of the bladder condition at that moment. Improvement is defined as a reduction in the number and/or severity of observed problems.
Time Frame: 12 Weeks (Randomized Phase) and 12 Months (Open Label Phase)
Population: Intent to Treat
Measure: Number; unit: percentage of patients that improved
Groups:
- Open Label Sham Treatement Group: Patients received active treatment with the VERV™ System for up to 9 additional months as part of the open label phase of the study.
Arm/Group | Active Treatment Group | Sham Treatment Group | Open Label Active Treatment Group | Open Label Sham Treatement Group
Number analyzed (Participants) | 80 | 83 | 15 | 18
percentage of patients that improved | 53.7 | 44.2 | 60.0 | 64.3
Statistical Analysis 1: Comparison: Active Treatment Group vs Sham Treatment Group; Test type: Superiority or Other; p = 0.4147, Fisher Exact
Statistical Analysis 2: Comparison: Open Label Active Treatment Group vs Open Label Sham Treatement Group; Test type: Superiority or Other; p = 0.0877, Fisher Exact

8. Secondary Outcome: Assessment of Treatment Benefit Scale (TBS)
Description: TBS is a patient-reported outcome comprised of a 4-point scale of checkboxes to describe the change in condition during treatment (greatly improved to worsened). Improvement was defined as a change in the patient's assessment of overall condition to improved or greatly improved over the course of treatment. Analysis was based upon the number of patients who reported an improvement in condition.
Time Frame: 12 Weeks
Population: Intent to Treat
Measure: Number; unit: percentage patients improved (responded)
Arm/Group | Active Treatment Group | Sham Treatment Group
Number analyzed (Participants) | 56 | 66
percentage patients improved (responded) | 55.4 | 42.4
Statistical Analysis 1: Comparison: Active Treatment Group vs Sham Treatment Group; Test type: Superiority or Other; p = 0.2032, Fisher Exact

9. Secondary Outcome: Assessment of Improvement as Measure by Overactive Bladder Satisfaction With Treatment Questionnaire (OAB-SAT)
Description: Overall satisfaction with treatment was assessed (OAB-SAT-q) an 11 question list with multiple scaled checkboxes to allow the subject to rate the treatment with regard to satisfaction, bother from side effects, treatment endorsement, and convenience.
Time Frame: 12 weeks
Population: Intent to treat population for those who had prior treatment for OAB.
Measure: Number; unit: percentage of patient prefer treatment
Arm/Group | Active Treatment Group | Sham Treatment Group
Number analyzed (Participants) | 32 | 34
percentage of patient prefer treatment | 65.3 | 57.6
Statistical Analysis 1: Comparison: Active Treatment Group vs Sham Treatment Group; Test type: Superiority or Other; p = 0.4151, Wilcoxon (Mann-Whitney) — Calculated for only those patients who had prior OAB treatment only

10. Secondary Outcome: Change Clinical Global Impressions at 12 Weeks
Description: CGI is an Investigator assessment, which rates the severity of illness at baseline on a scale of 1 (normal, not ill at all) to 7 (Amongst the most extremely ill patients), and then rates improvement at 12 weeks on a scale of 1 (very much improved) to 10 (very much worse). The analysis was based upon the number of patients that "much" and "very much" improved.
Time Frame: 12 weeks (Randomized Phase) and 12 Months (Open Label Phase)
Population: Intent to treat
Measure: Number; unit: % patients much or very much improved
Arm/Group | Active Treatment Group | Sham Treatment Group | Open Label Active Treatment Group | Open Label Sham Treatment Group
Number analyzed (Participants) | 80 | 83 | 9 | 13
% patients much or very much improved | 23.2 | 24.2 | 36.0 | 46.5
Statistical Analysis 1: Comparison: Active Treatment Group vs Sham Treatment Group; Endpoint defined as percentage of patients that "much improved" or "very much improved" following treatment; Test type: Superiority or Other; p = 0.9814, Fisher Exact
Statistical Analysis 2: Comparison: Open Label Active Treatment Group vs Open Label Sham Treatment Group; Test type: Superiority or Other; p = 0.7305, Fisher Exact

11. Primary Outcome: Evaluate the Median Change From Baseline in Mean Urgency (Urinary) Incontinence Episodes (Leaks) Between the Active and Sham Treatment Groups
Description: The primary objective of the randomized phase of the study is to evaluate the 12 week and 12 month median change from baseline in mean urgency (urinary) incontinence episodes (leaks) between treatment groups. The mean of the number of urinary incontinence episodes over 24 hours" is defined as the mean of the number of UIEs recorded per 24 hour period for three consecutive days (via a 3-day diary).
  Mean urinary frequency episodes calculated for each patient during time period. The median change in frequency was then calculated for each treatment group. Distribution of changes from baseline were then assessed prospectively for normality using the Kolmogorov - Smirnoff test. Since departure from normality was actually observed in the distribution, the Wilcoxon Rank-Sum test was performed to compare the median change between treatment groups and the p-values for the test of equality of medians were reported along with the medians.
Time Frame: 12 weeks (Randomized Phase) and 12 Months (Open Label)
Measure: Median (Inter-Quartile Range); unit: Episodes/day
Arm/Group | Active Treatment Group | Sham Treatment Group | Open Label Active Treatment Group | Open Label Sham Treatment Group
Number analyzed (Participants) | 68 | 75 | 25 | 26
Episodes/day | -3.7 [-4.7 to -1.0] | -1.7 [-3.3 to -1.0] | -1.2 [-3.2 to -0.3] | -1.0 [-2.3 to -0.3]
Statistical Analysis 1: Comparison: Active Treatment Group vs Sham Treatment Group; Test type: Superiority or Other; p = 0.2191, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Open Label Active Treatment Group vs Open Label Sham Treatment Group; Test type: Superiority or Other; p = 0.5357, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse Events reported over the course of 12 month treatment.
Description: 80 Active Treatment and 82 Sham patients included in analysis; 1 Sham patient withdrew on Day 1 prior to device placement and was excluded.
Groups:
- Randomized Active Treatment Group: VERV™ System
  (VERV™ System): Active electrode patches are worn for 12 weeks, one per week. The patch is placed by the subject. All subjects will have access to active patches for 9 months after the sham-controlled 12-week portion of the study is complete.
- Randomized Sham Treatment Group: Sham version of (VERV™ System)
  Sham version of (VERV™ System): Inactive (sham) electrode patches are worn for 12 weeks, one per week. The patch is placed by the subject. All subjects will have access to active patches for 9 months after the sham-controlled 12-week portion of the study is complete.
- Open Label Active Treatment Group; Open Label Sham Treatment Group: VERV™ System
  (VERV™ System): Active electrode patches are worn for up to 9 additional months, one per week during the open label phase.
Arm/Group | Randomized Active Treatment Group | Randomized Sham Treatment Group | Open Label Active Treatment Group | Open Label Sham Treatment Group
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/82 | 0/57 | 1/66
Other Adverse Events (participants affected / at risk) | 30/80 | 29/82 | 13/57 | 12/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Active Treatment Group (N=80) | Randomized Sham Treatment Group (N=82) | Open Label Active Treatment Group (N=57) | Open Label Sham Treatment Group (N=66)
Heart Attack (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Event not considered related to procedure or treatment.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Active Treatment Group (N=80) | Randomized Sham Treatment Group (N=82) | Open Label Active Treatment Group (N=57) | Open Label Sham Treatment Group (N=66)
Skin Irritation (Injury, poisoning and procedural complications) | 12 (17) | 5 (6) | 5 (8) | 12 (27) — redness,erythema, itching, irritation, blistering
Change in Bowel Habit (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) — Diarrhea
Urinary Tract Infection (Infections and infestations) | 1 (1) | 2 (2) | 2 (4) | 0 (0) — UTI
Redness and Itchiness (Injury, poisoning and procedural complications) | 18 (26) | 12 (18) | 7 (10) | 11 (18) — Redness/erythema and itchiness
Rash (Injury, poisoning and procedural complications) | 7 (9) | 6 (9) | 6 (6) | 7 (9) — Rash
Blistering (Injury, poisoning and procedural complications) | 2 (3) | 3 (4) | 2 (2) | 1 (1) — Blisters
Allergic Reaction to Sulfa (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Allergic Reaction
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5) | 1 (1) | 2 (2)
Chest Pain/Shortness of Breath (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cold/Flu (Infections and infestations) | 2 (2) | 3 (3) | 1 (1) | 1 (1)
Environmental Allergies (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea/Vomiting due to Food Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Kidney/Ureteral Stones and bleedling (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Foot Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sleeping Difficulties (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Burning sensation at Patch Site (Injury, poisoning and procedural complications) | 1 (1) | 2 (3) | 2 (2) | 2 (3) — Sensory
Pain at Patch Site (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Sensory
Numbness (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 0 (0) — Sensory
Tingling Sensation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Sensory

LIMITATIONS AND CAVEATS:
There was a higher than anticipated rate of patient withdrawals observed in both groups due to skin irritation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No